CLINICAL TRIAL: NCT05563051
Title: Kaneka Endovascular Embolization and Protection
Acronym: KEEP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kaneka Medical America LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KMA-IVRNV-001
Record Dates: First submitted 2022-09-28; First posted 2022-10-03 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Aneurysm Cerebral
Keywords: aneurysm; coil; i-ED COIL; embolization; neuro endovascular
MeSH Terms: conditions — Intracranial Aneurysm; Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Interventional treatment (Other): Open label
  Interventions: Device: i-ED COIL

INTERVENTIONS:
Device: i-ED COIL — The i-ED COIL System (i-ED COIL and detachment box) are intended for the endovascular embolization of intracranial aneurysms and other neurovascular abnormalities such as arteriovenous malformations and arteriovenous fistulae.
  Other Names: Embolic coils; Embolization coils

SUMMARY:
Prospective, multi-center, non-randomized registry / study, up to 164 patients enrolled and followed at 180 days +/- 45 days and again at 365 days +/- 90 days post procedure

DETAILED DESCRIPTION:
Assess and describe real world clinical data on i-ED coils Characterize the acute and long-term performance of iED coils when used for treating for an intracranial aneurysm May be used alone or in combination with other adjunctive device(s)

Study Duration

Anticipated timeline for study:

Patient enrollment in 18 - 24 months Completion of follow-up 12 months after last patient enrolled

ELIGIBILITY:
Inclusion Criteria:

* Target aneurysm of 4mm - 14mm in size
* Ruptured or unruptured
* Suitable for embolization with coils
* May be treated with or without assist devices

Exclusion Criteria:

* Unstable neurological deficit in unruptured cases (condition worsening within last 90 days)
* Pre-planned staged procedure of target aneurysm
* mRS score 3 or more
* Hunt Hess Score more than 3 for subjects with ruptured aneurysm
* Evidence of active infection (e.g.,fever, temperature >38 degrees C and/or WBC >15,000)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2022-12-13 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Adequate Occlusion | 12 months
  Proportion of subjects who achieve Adequate Occlusion (Modified Raymond-Roy I or II Classification)

SECONDARY OUTCOMES:
Complete Occlusion | 12 months
  Complete occlusion at 1 year (Modified Raymond-Roy I)
Packing Density | 12 months
  Aneurysm volume and percent of aneurysm packing for coil embolization. Packing density will be evaluated based on aneurysm volume and coil volume
Modified Rankin Score | 12 months
  Modified Rankin Score (Scale from 0-6), the lower the score the better - 0 No symptoms and 6 is dead.
  1. No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. Slight disability. Able to look after own affairs without assistance but unable to carry out all previous activities.
  3. Moderate disability. Requires some help, but able to walk unassisted.
  4. Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. Dead
Retreatment | 12 months
  Any retreatment of the aneurysm, surgically or interventional embolization
Adverse events | 12 months
  Device or procedure related adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Ajit Puri, MD, Principal Investigator — University of Massachusetts, Worcester; Mohamed Hussain, MD, Principal Investigator — The Cleveland Clinic
Locations (4):
- United States (4):
  - McLaren Health Care, Grand Blanc, Michigan
  - Northwell Health Lenox Hill Hospital, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - SSM Health St. Anthony's Hospital, Oklahoma City, Oklahoma

IPD SHARING:
Plan to Share IPD: No